CLINICAL TRIAL: NCT02694263
Title: A Randomised Controlled Trial for People With Established Type 2 Diabetes During Ramadan: Canagliflozin (Invokana™) vs. Standard Dual Therapy Regimen: The 'Can Do Ramadan' Study
Brief Title: Canagliflozin (Invokana™) vs. Standard Dual Therapy Regimen for T2DM During Ramadan
Acronym: Can Do
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0527
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; repaglinide; Pioglitazone; Gliclazide; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Canagliflozin + Metformin (Experimental): Canagliflozin + metformin (using the participant's current dose, or dose recommended by the study clinician). An initial dose of 100mg once daily of Canagliflozin will be prescribed, and this will be titrated up to a maximum of 300mg once daily.
  Interventions: Drug: Canagliflozin
- Repaglinide + Metformin (Active Comparator): Repaglinide + Metformin (using the participant's current dose(s), or dose recommended by the study clinician). An initial dose of 0.5mg once daily where no prior treatment has been given will be prescribed. However, where prior treatment has been in place, an initial dose of 1-2mg once daily will be started and this will be titrated up to a maximum dose of 4mg daily.
  Interventions: Drug: Repaglinide
- Pioglitazone + Metformin (Active Comparator): Piogliazone + Metformin (using the participant's current dose(s), or dose recommended by the study clinician). For example, Pioglitazone dose will initially be 15mg or 30mg once daily. If the response is inadequate, the maximum daily dosage will be increased to 45mg once daily.
  Interventions: Drug: Pioglitazone
- Gliclazide + Metformin (Active Comparator): Gliclazide + Metformin (using the participant's current dose(s), or dose recommended by the study clinician). For example, Gliclazide dose will initially be 40-80 mg once daily, up to maximum dose of 160mg twice daily..
  Interventions: Drug: Gliclazide
- Glimepiride + Metformin (Active Comparator): Glimepiride + Metformin (using the participant's current dose(s), or dose recommended by the study clinician). Glimepiride will initially be administered as 1mg once daily, up to a maximum dose of 4mg once daily.
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Canagliflozin — Comparison of Canagliflozin (Invokana™) vs. standard dual therapy (Repaglinide, Pioglitazone, Gliclazide or Glimepiride) for the treatment of Type 2 Diabetes.
  Other Names: Invokana
  Arms: Canagliflozin + Metformin
Drug: Repaglinide — Comparison of Canagliflozin (Invokana™) vs. standard dual therapy (Repaglinide) for the treatment of Type 2 Diabetes.
  Other Names: Prandin
  Arms: Repaglinide + Metformin
Drug: Pioglitazone — Comparison of Canagliflozin (Invokana™) vs. standard dual therapy (Pioglitazone) for the treatment of Type 2 Diabetes.
  Other Names: Actos
  Arms: Pioglitazone + Metformin
Drug: Gliclazide — Comparison of Canagliflozin (Invokana™) vs. standard dual therapy (Gliclazide) for the treatment of Type 2 Diabetes.
  Other Names: Diamicron
  Arms: Gliclazide + Metformin
Drug: Glimepiride — Comparison of Canagliflozin (Invokana™) vs. standard dual therapy (Glimepiride) for the treatment of Type 2 Diabetes.
  Other Names: Amaryl
  Arms: Glimepiride + Metformin

SUMMARY:
This study aims to determine if the addition of Canagliflozin (Invokana™) therapy to monotherapy of metformin is more effective at achieving the double composite endpoint of a reduction in HbA1c (≥ 0.3%) and weight loss (≥1kg) 3-4 weeks post-Ramadan. The study will also include patients currently on dual therapy, specifically metformin plus a sulphonylurea, pioglitazone or repaglinide to determine whether switching to metformin plus Canagliflozin (Invokana™) is more effective at achieving the composite endpoint compared to those remaining on previous dual therapy. There are a number of secondary outcomes including weight loss, rates of hypoglycaemia, blood pressure and a number of biochemical endpoints.

DETAILED DESCRIPTION:
There are over one billion Muslims in the world with the majority participating in Ramadan. The prevalence of diabetes in several countries with large Muslim populations is similar to the rates observed in westernised countries, which increases by 10% annually as a result of urbanization and socioeconomic development. Observance of Ramadan is an integral part of Islamic identity being one of the five main pillars that constitute this widely followed religion. Muslims observing Ramadan are required to fast from sunrise to sunset during this holy month. The timing of Ramadan follows the lunar calendar which occurs 10 days earlier each year; this means that the fasting period coincides with the summer season for many consecutive years before moving in line with the winter months. During the summer season Ramadan can take place with the longest hours of daylight which has a greater impact and risk for people with diabetes who fast during this period.

Although the Quran exempts "sick" people from the duty of fasting many Muslims with diabetes do not consider themselves to be sick and are keen to fast. A recent epidemiological study involving 13 Islamic countries reported that 43% of patients with Type 1 diabetes mellitus (T1DM) and 79% of people with type 2 diabetes mellitus (T2DM) fast during this religious period.

Concern for Muslims with diabetes fasting during Ramadan has been recognised by religious leaders and indeed 2009 saw a landmark event. A statement was issued at the meeting of the Council of the International Islamic Fiqh Academy of the Organisation of Islamic Conference at its 19th session. In brief, people with diabetes were classified into four categories in line with expert recommendations published in 2005. Categories 1 and 2 include those with diabetes at very high risk of serious complications and high risk of complications due to fasting, respectively. These two groups are exempt from observing Ramadan. Categories 3 and 4 include those with diabetes who have a medium risk of complications and those with a low risk of complications due to fasting, respectively. The latter two groups are not automatically exempt from observing Ramadan. The risk of complications in this context refers specifically to the likelihood of hypoglycaemic events, and includes other acute illnesses associated with diabetes, patients on renal dialysis, women with diabetes during pregnancy, patients with macrovascular disease, and those who live alone and are on insulin therapy or oral insulin secretagogues. Additionally, all people with T1DM are classed as category 1. However, the impact of the feasting part of Ramadan, for example on hyperglycaemia or deterioration of glycaemic control, is not considered in this statement. Furthermore, it is not known to what extent these guidelines are followed in practice.

There is an abundance of evidence describing the impact of Ramadan on people with T2DM from retrospective to population-based studies. However, there is a lack of evidence available to help guide the management of people with diabetes who wish to observe Ramadan. Fasting and feasting during this holy month can cause health risks for people with diabetes. The Epidemiology of Diabetes and Ramadan 1422/2001 Study ("EPIDAR") was a large population-based, international epidemiological study of diabetes conducted in 13 countries with Muslim populations. One of the aims of this study was to determine the potential effects of fasting in people with diabetes on their well-being and the management of this condition. They observed a 7.5-fold (from 0.4 to 3 events per 100 per month) increased risk of severe hypoglycaemia in patients with T2DM as a result of a change in eating patterns during Ramadan. Severe hypoglycaemia was defined as hypoglycaemia leading to hospitalization. Additionally a 5-fold increase in the incidence of severe hyperglycaemia with/without ketoacidosis was observed in patients with T2DM.

Other risks for people with diabetes who fast during Ramadan include diabetic ketoacidosis due to a lack of insulin, dehydration due to lack of fluid intake during the fasting period, and orthostatic hypotension in addition to an increased risk of thrombosis due to increased blood viscosity secondary to dehydration. Only 62% of those with T2DM in the "EIPDAR" study reported receiving recommendations from their health care providers. These recommendations should include changes in lifestyle (diet and physical activity) and in medication choice and dosage to limit the potential complications of fasting and feasting for this patient population.

There have been significant advances in glucose lowering therapies in T2DM and their availability, thus offering a greater choice of therapies to people with diabetes with the potential for supporting safer fasting. Three new classes of therapy have been licensed for the treatment of T2DM in the United Kingdom (UK) in the past 10 years. The most recent class that has been introduced are the Sodium Glucose Co-Transporter 2 Inhibitors (SGLT2 inhibitors). There are six known members of the SGLT family to date. Canagliflozin (Invokana™), a once daily tablet, is one of a number of SGLT2 inhibitors that have been licensed within the UK. This medication is taken once daily orally (either 100 or 300mg). Phase III trials of this novel agent have reported reductions in HbA1c between 0.70 and 1.16%, body weight reduction between 1.8 and 3.7% and systolic blood pressure reduction between 1.6 and 6.6mmHg (millimetre of mercury) from baseline. Canagliflozin (Invokana™) has a low intrinsic propensity to cause hypoglycaemia. Importantly this drug is reported to be well-tolerated and has a good safety profile in patients with inadequately controlled T2DM as monotherapy or in combination with other glucose lowering therapy including sulphonylureas and metformin.

In 2016, Ramadan takes place throughout the months of June and July. At this time of year in the UK, between dawn and sunset there are approximately 14.5 hours of daylight at the beginning and 13 hours towards the end of Ramadan during which there is fasting. This is a significant portion of the 24 hour day; thus abstinence from food for such a prolonged period poses an increased risk for those with T2DM especially if their medicine regimens are not altered to accommodate this. In light of this the study aims to determine if the addition of Canagliflozin (Invokana™) therapy to monotherapy of metformin is more effective at achieving the double composite endpoint of a reduction in HbA1c (≥ 0.3%) and weight loss (≥1kg) 3-4 weeks post-Ramadan. The study will also include patients currently on dual therapy, specifically metformin plus a sulphonylurea, pioglitazone or repaglinide to determine whether switching to metformin plus Canagliflozin (Invokana™) is more effective at achieving the composite endpoint compared to those remaining on previous dual therapy. There are a number of secondary outcomes including weight loss, rates of hypoglycaemia, blood pressure and a number of biochemical endpoints.

The study will also include an objective measure of glycaemic status using a Flash Glucose Monitoring System (FGMS) called a "FreeStyle Libre" sensor in a sub-set of participants (15-20 participants). Participants can 'opt-in' to the FGMS sub-study and the device will be worn before medication is initiated and at the first follow-up visit 3-4 weeks post Ramadan. The study will also invite those participating in the sub-study to wear the device during Ramadan. The use of FGMS will provide up to 14 days of blood glucose readings taken every 15 minutes allowing us to apply glycaemic thresholds to the uploaded data and calculate the proportion of time spent in hypo, hyper or normoglycaemic states in the two treatment groups.

There is limited evidence on the changes in levels of physical activity for people who observe Ramadan. It is widely believed that levels of physical activity are reduced due to a fear of feeling too weak [29]. To address this, the study will objectively measure physical activity levels before, during and after Ramadan in a sub-set of participants (15-20 participants) in addition to using the self-reported validated international physical activity questionnaire (IPAQ).

It is hypothesised that therapy based on Canagliflozin (Invokana™) is more effective than sulphonylurea-based regimen at helping people with established T2DM who are observing Ramadan to achieve the double composite endpoint of a reduction in HbA1c (≥ 0.3%) and weight loss (≥1kg) 3-4 weeks post-Ramadan.

STUDY DESIGN

This is an open label randomised controlled trial with two cohorts:

1. Cohort 1 - Individuals on metformin monotherapy will be randomised (1:1) to either the addition of Canagliflozin (Invokana™) or repaglinide, a sulphonylurea or pioglitazone, and
2. Cohort 2 - Individuals on dual therapy (metformin plus repaglinide, a sulphonylurea or pioglitazone) will be randomised (1:1) to either continuation of their current therapy or to switch to metformin and Canagliflozin (Invokana™) Randomisation will be stratified by site and entry therapy (monotherapy OR dual therapy which includes metformin plus pioglitazone, or metformin plus either a sulphonylurea or repaglinide, respectively) resulting in 6 stratification groups. Randomisation will not be carried out until after the baseline data have been collected.

The intervention group in Cohort 1 will be those randomised to metformin + Canagliflozin (Invokana™). The control group in Cohort 1 will be those randomised to receive metformin plus repaglinide, or a sulphonylurea or pioglitazone in line with current National Institute for Health and Care Excellence (NICE) guidance as the preferred second-line therapy after metformin.

The intervention group in Cohort 2 will be those randomised to switch to metformin plus Canagliflozin (Invokana™). The control group in Cohort 2 will be those who continue with their current medication.

The study will recruit patients from both primary and secondary care in Leicester and Birmingham. It is envisaged to commence recruitment in February 2016, although this date is conditional upon on ethics committee and regulatory approval and necessary preparatory arrangements, including research governance approval at both sites. Actively recruitment will begin once all approvals are in place and after Sponsor 'green light' has been issued.

Randomisation and Code breaking:- There will be six randomisation lists. Participant identifier numbers will be assigned sequentially as each subject enters the study. The participant will be assigned a study drug through a randomisation schedule based on the randomisation plan.

Randomisation will be stratified by site and entry therapy (monotherapy OR dual therapy which includes metformin plus pioglitazone or metformin plus either a sulphonylurea or repaglinide) resulting in 6 groups using a variable block size of between 4 and 6. Participants will be randomised 1:1 to metformin + Canagliflozin (Invokana™) or to metformin + a sulphonylurea, or continuation of their sulphonylurea, repaglinide or pioglitazone.

Discontinuation/Withdrawal of Participants from Study Treatment:- Each participant has the right to withdraw from the study at any time without giving a reason and without any future care being affected. The investigator may discontinue a participant from the study at any time if the investigator considers it necessary for any reason. The reason for withdrawal will be recorded in the case report form (CRF) and documented in the medical notes. If the participant is withdrawn due to an adverse event, the Investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved, stabilised or concluded.

Source Data:- Source documents are original documents, data, and records from which participants' CRF data are obtained. These include, but are not limited to, hospital records (from which medical history and previous and concurrent medication may be summarised into the CRF), clinical and office charts, laboratory and pharmacy records, diaries, microfiches, radiographs, and correspondence. CRF entries will be considered source data if the CRF is the site of the original recording (e.g., there is no other written or electronic record of data). Specifically, for this study the CRF will be used as the source document for all anthropometrics, questionnaire and biochemistry that is collected during the study visits and copy of the biochemistry and anthropometric results will be put into the patient medical notes.

Drug Management Storage of Study Treatment:- The local National Health Service (NHS) Trust pharmacies will supply the licensed products and will handle it according to their in-house protocols. The study will be conducted in accordance with the Helsinki declaration. All staff working on this study will have an up to date International Council for Harmonisation -Good Clinical Practice (ICH-GCP) certificate.

Compliance with Study Treatment:- The study will measure compliance by requesting participants to bring all unused or part-used medications and packaging from used medication at each visit. This will be recorded in the drug accountability log as part of the CRF. A participant who ceases to take their medication for up to two weeks will be considered 'non-compliant'. They will have the opportunity to re-initiate medication.

Accountability of the Study Treatment:- The local NHS Trust pharmacies will dispense the study medication from their own stocks and they will also provide the appropriate drug labels. Returned and unused medication will be recorded by the research team and the research team will provide pharmacy with this medication at the end of the visit so that they can be destroyed in accordance with local regulations. Metformin will be prescribed as per usual by their General Practitioner (GP).

Concomitant Medication:- Throughout the study, Investigators may prescribe any concomitant medications or treatments deemed necessary to provide adequate supportive care except for those listed in the exclusion criteria. If the participant is subsequently prescribed excluded medication they will be withdrawn from the study.

SAFETY REPORTING Please note the Sponsor of the Study (University of Leicester) and the Chief Investigator shall be responsible for complying with UK Competent Authority (Medicines and Healthcare products Regulatory Agency (MHRA)) safety reporting requirements and be responsible for the participating (co- or sub-) investigators, as defined in the applicable laws and regulations.

As provided for in Article 3 of the Research Funding Agreement, the Sponsor and Chief Investigator will submit the safety information requested on the 'Clinical Serious Adverse Event Report' form (FRM-09210, Version 9.0) to the identified Janssen Pharmaceuticals Inc. representative of the country of origin, (i.e., Drug Safety Department of Janssen-Cilag Ltd) either by fax 01494 567799, or secure email and pdf to "Dsafety@its.jnj.com". For additional support, the Janssen-Cilag Ltd Drug Safety Department can be contacted on 01494 567 447.

Reporting Procedures for All Adverse Events (AEs):- All AEs occurring during the study observed by the investigator or reported by the participant, whether or not attributed to study medication, will be recorded on the CRF. The following information will be recorded, description, date of onset and end date, severity, assessment of relatedness to study medication, other suspect drug or device and action taken. Follow-up information will be provided as necessary.

Reporting Procedures for Serious Adverse Events (SAEs):- All SAEs must be reported to the Sponsor within one working day of discovery or notification of the event. The Sponsor will perform an initial check of the information and ensure that it is reviewed at the next R&D Management meeting. All SAE information must be recorded on an SAE form and sent to the Sponsor. Additional information received for a case (follow-up or corrections to the original case) needs to be detailed on a new SAE form and sent to the Sponsor.

The Sponsor will report all Suspected Unexpected Serious Adverse Reactions (SUSARs) to the MHRA and the Research Ethics Committee (REC) concerned. Fatal or life-threatening SUSARs must be reported within 7 days and all other SUSARs within 15 days. The Chief Investigator will inform all investigators concerned of relevant information about SUSARs that could adversely affect the safety of participants. The Sponsor will use the Summary of Product Characteristics (SMPC) as the Reference Safety Information (RSI) when determining the expectedness of any untoward medical occurrences and thus SAE/SUSAR reporting.

In addition to the expedited reporting above, the Chief Investigator will submit once a year throughout the clinical study or on request a Development Safety Update Report (DSUR) to the MHRA and REC.

STATISTICS Description of Statistical Methods:- Participants recruited to the study will be compared by randomised group with respect to both their baseline characteristics and their pre-Ramadan characteristics. Numbers (with percentages) for binary and categorical variables and means (and standard deviations), or medians (with lower and upper quartiles) for continuous variables will be presented. There will be no tests of statistical significance nor confidence intervals for differences between randomised groups on any baseline variable.

The primary outcome of this study is the achievement of the double composite endpoint of a reduction in HbA1c (≥ 0.3%) and weight loss (≥1kg) 3-4 weeks post-Ramadan.

All analyses of outcome data will be carried out on a complete case basis according to randomised group. As a sensitivity analysis, for the primary and main secondary outcome, multiple imputations will be used to perform an intention to treat analysis. The investigator will also conduct a per protocol analysis excluding those who report no longer taking their randomised treatment at the two follow-ups. All analyses will be performed assessing change during the following time periods:

* Baseline to 3-4 post-Ramadan data constituting the primary analysis
* Pre-Ramadan to 3-4 weeks post-Ramadan ±2 weeks
* Baseline to 12 weeks post-Ramadan ±2 weeks
* Baseline to 12 months post-baseline ±6 weeks The primary outcome will be analysed using logistic regression adjusted for the stratification factors (site, entry therapy ((1) monotherapy (2) dual therapy metformin plus pioglitazone (3) dual therapy metformin plus either a sulphonylurea or repaglinide)). The dependent variable will be defined as those achieving all of the composite end point targets. The same analysis method will be used for the secondary composite outcomes.

The biomedical outcomes will be analysed using linear regression adjusted for the stratification factors and baseline value. Ordinal regression will be used to compare treatment groups for the treatment satisfaction scores. Linear regression will be used for total metabolic equivalent (total METs).

The percentage of patients experiencing one or more self-reported hypoglycaemic events in their diaries (defined as a blood glucose level of ≤3.9 mmol/l) will be reported by group along with the median (Inter Quartile Range) number of episodes per patient. The incidence rate of hypoglycaemia per person year will be calculated per group and compared using the incidence rate ratio (IRR).

Continuous Glucose Monitoring System (CGMS) data will be collected at 3 time points. The mean proportion (%) of time spent either above (≥10mmol/l), below (≤3.1mmol/l) or within (3.2-9.9mmol/l) - which are our predefined glycaemic ranges - will be calculated for each participant over the recording period and adjusted for 24 hours. The study will compare these by treatment group for each time-point. The investigator will calculate change in proportion of time spent in each category from pre-Ramadan against during and against post-Ramadan within each group. The investigator will then compare any identified glycaemic shifts between treatment groups. The investigator will calculate the number of Continuous Glucose Monitor (CGM) low glucose events (≤3.1 and ≤2.2mmol/L) and CGM high glucose events (≥10.0mmol/L) within each treatment group and determine if the incidence changes across the three time points.

The Number of Participants:- The sample size required to detect a minimum clinical significant difference of 27.7% in those achieving the primary outcome between the treatment arms is 116 participants (n=58 per group), with 80% power and an alpha of 5%, assuming a dropout rate of 20%. This is based on 21.2% of the SU plus metformin group in the 'Treat 4 Ramadan study' having met the proposed primary outcome of achieving the double composite endpoint of a reduction in HbA1c (≥0.3%) and weight loss (≥ 1kg) 3-4 weeks post-Ramadan.

The Level of Statistical Significance:- All analyses will be carried out in Stata (version 12.0) 95% confidence intervals will be reported with p<0.05 relating to statistical significance.

Procedure for Accounting for Missing, Unused, and Spurious Data:- Data will be entered into a database with real-time validation, which will limit spurious data. Before analysis begins all data will be checked and any anomalies will be checked against the source data.

During data collection the study team will attempt to minimise missing data items. Participants with missing data will be excluded on a case-wise basis, i.e., only from those analyses which required the missing items. The primary and main secondary outcomes will be analysed on both a complete case basis and using multiple imputation to estimate the effect of missing data.

QUALITY CONTROL AND QUALITY ASSURANCE PROCEDURES A monitoring plan will be developed by the Sponsor in accordance with Sponsor Standard Operating Procedures (SOPs). The monitoring plan will be based on a study risk assessment which is determined by the level of risk within the study to participant safety and data integrity and validity; monitoring will be carried out by monitoring staff employed by the Sponsor.

The Leicester Diabetes Centre in conjunction with the Leicester Clinical Trials Unit will be responsible for all elements of study management on an ongoing basis. For example, the CRFs will be checked for completeness at the end of a measurement session and any data queries will be raised with the research nurse who recorded the data in the first instance. Repeated errors will be referred to the Senior Research Team Manager who will instigate training. The study monitor will remain external to the study team thereby ensuring independence during the sponsor monitoring process. All in-house monitoring and audit will be performed by staff who are ICH/GCP trained and are competent in monitoring to GCP standards. A documented monitoring log and audit trail will be maintained throughout the lifetime of the study.

The Trial Manager in conjunction with the Clinical Trials Unit will oversee the set-up of and conduct of study procedures at each site. All source data, study documents, medical notes will be made available for Sponsor monitoring, and any external audits and inspections as appropriate, for example by the MHRA or Research Ethics Committee.

STUDY GOVERNANCE Trial Steering Committee (TSC):- TSC will comprise an independent chair, at least one other independent clinician with expertise in the management of diabetes, the chief investigator, key co-investigators, and representation from the Leicester Clinical Trials Unit. The study statisticians may attend as needed. This committee will be responsible for the overall management and oversight of the study and will meet once prior to start up and then every 6 months, normally within 2 months of the Data Safety Monitoring Committee (DSMC) (although additional meetings may be called by the Chief Investigator or TSC or DSMC chair) to review and approve protocol amendments and any sub-study proposals, review recruitment rates, protocol adherence, retention, compliance, safety issues, planned analyses and reports and act on recommendations of the DSMC. A copy of meeting minutes will be sent to the Sponsor.

Data Safety Monitoring Committee (DSMC):- DSMC will comprise an independent chair, independent clinician and independent statistician. The chief investigator or study statistician may be invited to attend to provide specific input by the DSMC Chair. The DSMC will be responsible for the interests and safety of the participants and its main role will be to make advisory recommendations to the TSC who will report to the Sponsor. To this end, the DSMC will undertake safety data reviews every six months after the first 5 participants are recruited unless otherwise deemed necessary. In addition, the DSMC will review analysis plans.

Project Management Committee (PMC):- PMC will report to the TSC and will include the chief investigator, other senior investigators and the day-to-day project management team. The group will meet monthly or bi-monthly depending on need, either face-to-face or by teleconference, to discuss the details and logistics of recruitment, retention and follow-up data collection.

ELIGIBILITY:
Inclusion Criteria

1. Able, in the opinion of the Investigator, and willing to give informed consent
2. Age ≥ 25 years old
3. Established T2DM (≥ 3 months) on stable dose monotherapy (metformin only for ≥ 8 weeks prior to enrolment) OR stable dose dual therapy (metformin plus either repaglinide, a sulphonylurea or pioglitazone or DPP-4 inhibitor for ≥ 8 weeks prior to enrolment)
4. HbA1c between 6.6 - 11% (49mmol/mol - 97mmol/mol) at the screening visit
5. Individuals intending to fast during the holy month of Ramadan

Exclusion Criteria

1. Unable, in the opinion of the Investigator, and unwilling to provide informed consent
2. Aged < 25 years old
3. Established T2DM (≤ 3 months) on medication for fewer than 8 weeks prior to enrolment
4. HbA1c ≤6.5 and ≥11.1%
5. Individuals not intending to fast during the holy month of Ramadan
6. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods. The latter includes avoiding sex, hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization, consistent with local regulations regarding use of birth control methods for subjects participating in clinical trials, for the duration of their participation in the study, or not heterosexually active. Furthermore, subjects who are not heterosexually active at screening must agree to utilize a highly effective method of birth control if they become heterosexually active during their participation in the study. Women of childbearing potential must have a negative urine pregnancy test at baseline.
7. Suffer from terminal illness
8. Have renal disease that requires immunosuppressive therapy, dialysis or transplant
9. Have nephrotic syndrome or inflammatory renal disease
10. Have an estimated glomerular filtration rate (eGFR) <60ml/min/1.73m2 at screening
11. Have serum creatinine levels >132.6μmol/L for men or >123.8μmol/L for women
12. Impaired liver function (ALAT ≥ 2.5 times upper limit of normal)
13. Known Hepatitis B antigen or Hepatitis C antibody positive
14. Clinically significant active cardiovascular disease (including history of myocardial infarction, unstable angina, previous revascularization procedure or cerebrovascular accident) within the past 6 months before screening
15. Have uncontrolled hypertension (defined as systolic blood pressure ≥180mm/Hg and diastolic ≥100mm/Hg in the supine position after >5minutes rest with confirmed compliance to antihypertensive medication)
16. Heart failure (NYHA class III and IV) at the discretion of the investigator
17. Previous history of recurrent major hypoglycaemia as judged by the study clinician
18. Known or suspected allergy to the study product
19. Receipt of any investigational drug within four weeks prior to this study
20. Has had previous treatment with a GLP-1 receptor agonist, insulin, or another SGLT2 inhibitor within 12 weeks of screening
21. Have severe and enduring mental health problems
22. Are not primarily responsible for their own care
23. Are receiving insulin therapy
24. Type 1 diabetes
25. Any contraindication to sulphonylureas, repaglinide, pioglitazone and/or DPP-4 inhibitors
26. Have severe irritable bowel disorder
27. Have hereditary glucose-galactose malabsorption
28. Have primary renal glycosuria
29. Patients who have participated in another study of an investigational medicinal product in the last 3 months
30. High risk of bone fracture (undiagnosed osteoporosis) as determined by the WHO FRAX tool
31. Evidence of excessive and compulsive drinking of alcohol i.e. alcohol abuse as determined by the Fast Alcohol Screening Test (FAST)
32. Individuals on a severe calorie restricted diet <800cals/day
33. Has a surgical procedure booked in the next 12 months
34. Has a history of chronic pancreatitis
35. Has latent autoimmune diabetes in adults (LADA)
36. Individuals on loop diuretics
37. Any contraindication to the IMP

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
HbA1c + weight loss | Baseline and 3-4 weeks post-Ramadan
  Double composite endpoint of a change in HbA1c (≥ 0.3%) and weight loss (≥1kg) between baseline and 3-4 weeks post-Ramadan.

SECONDARY OUTCOMES:
HbA1c + weight loss + Hypoglycaemic events | Baseline and 3-4 weeks post-Ramadan
  Triple composite endpoint of a reduction or maintenance of HbA1c, reduction in weight (≥ 1kg) and no hypoglycaemic events between baseline and 3-4 weeks post-Ramadan.
HbA1c | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in HbA1c level (%)
Fructosamine | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in Fructosamine
Body weight (kg) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in body weight (kg)
Systolic blood pressure (mm Hg) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in systolic blood pressure (mm Hg)
Diastolic blood pressure (mm Hg) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in diastolic blood pressure (mm Hg)
Total cholesterol (mmol/L) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in total cholesterol (mmol/L)
HDL cholesterol (mmol/L) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in HDL cholesterol (mmol/L)
LDL cholesterol (mmol/L) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in LDL cholesterol (mmol/L)
Triglycerides (mmol/L) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in Triglycerides (mmol/L)
Diabetes Treatment Satisfaction | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in Diabetes Treatment Satisfaction (DTSQ)
Physical Activity (self-reported) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in self-reported physical activity levels (measured using the International Physical Activity Questionnaire; IPAQ)
Physical Activity (GENEActiv) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in light, moderate, and vigorous intensity physical activity levels (measured using the GENEActiv device)
Hypoglycaemic events (change) (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in frequency of self-measured and self-reported hypoglycaemic events
Severe hypoglycaemic events (change) (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Mean change in frequency of self-measured and self-reported severe hypoglycaemic events
Hypoglycaemic events (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Median (interquartile range; IQR) number of self-measured and self-reported hypoglycaemic events per patient
Severe hypoglycaemic events (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Median (interquartile range; IQR) number of self-measured and self-reported severe hypoglycaemic events per patient
Hypoglycaemic events (per person year) (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Incidence rate of self-measured and self-reported hypoglycaemic events per person year (incidence rate ration; IRR).
Severe hypoglycaemic events (per person year) (self-measured) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Incidence rate of self-measured and self-reported severe hypoglycaemic events per person year (incidence rate ration; IRR).
Weight loss (kg) + severe hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of weight loss (kg) and no severe hypoglycaemic events.
No weight gain (kg) + reduction of hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of no weight gain (kg) and a reduction in the number of self-measured and self-reported hypoglycaemic events (+/- symptoms).
HbA1c (%) + severe hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of improved HbA1c (%) and no self-measured and self-reported severe hypoglycaemic events.
HbA1c (%) + hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of improved HbA1c (%) and a reduction in the number of self-measured and self-reported hypoglycaemic events.
No weight gain (kg) + HbA1c (%) | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of no weight gain (kg) and improved HbA1c (%).
No weight gain (kg) + severe hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of no weight gain (kg) and no self-measured and self-reported severe hypoglycaemic events.
No weight gain (kg) + no hypoglycaemic events | Baseline and (a) 3-4 weeks post-Ramadan, (b) 12 weeks post-Ramadan and (c) 12 months post-Ramadan.
  Double composite endpoint of no weight gain (kg) and no self-measured and self-reported hypoglycaemic events.
Hospital admissions | Beginning and end of Ramadan (i.e., during the month of Ramadan)
  Comparison of the number of hospital admissions between groups for complications related to diabetes during Ramadan.
Flash Glucose Monitoring - Time in glycaemic range | Baseline and (a) 3-4 weeks post-Ramadan, and (b) during Ramadan.
  Change in proportion of time spent in each glycaemic range (measured using the Flash Glucose Monitoring (FGM) device) calculated between treatment groups.
Flash Glucose Monitoring - Incidence | Baseline and (a) 3-4 weeks post-Ramadan, and (b) during Ramadan.
  Incidence of hypoglycaemic events and severe hypoglycaemic events (measured using the Flash Glucose Monitoring (FGM) device).
Flash Glucose Monitoring - Change | Baseline and (a) 3-4 weeks post-Ramadan, and (b) during Ramadan.
  Change in the frequency of hypoglycaemic events and severe hypoglycaemic events (measured using the Flash Glucose Monitoring (FGM) device).
Flash Glucose Monitoring - MAGE | Baseline and (a) 3-4 weeks post-Ramadan, and (b) during Ramadan.
  Change in the mean average glucose excursion (MAGE; measured using the Flash Glucose Monitoring (FGM) device).

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MBBS MD FRCP FRCGP, Principal Investigator — University of Leicester; Wasim Hanif, MBBS MD FRCP, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available. Abnormal blood results will be shared with the participant's general practitioner (GP) if it is considered to the clinically necessary.

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Salti I, Benard E, Detournay B, Bianchi-Biscay M, Le Brigand C, Voinet C, Jabbar A; EPIDIAR study group. A population-based study of diabetes and its characteristics during the fasting month of Ramadan in 13 countries: results of the epidemiology of diabetes and Ramadan 1422/2001 (EPIDIAR) study. Diabetes Care. 2004 Oct;27(10):2306-11. doi: 10.2337/diacare.27.10.2306. PMID 15451892
- [Background] Al-Arouj M, Bouguerra R, Buse J, Hafez S, Hassanein M, Ibrahim MA, Ismail-Beigi F, El-Kebbi I, Khatib O, Kishawi S, Al-Madani A, Mishal AA, Al-Maskari M, Nakhi AB, Al-Rubean K. Recommendations for management of diabetes during Ramadan. Diabetes Care. 2005 Sep;28(9):2305-11. doi: 10.2337/diacare.28.9.2305. No abstract available. PMID 16123509
- [Background] Li H, Gu Y, Zhang Y, Lucas MJ, Wang Y. High glucose levels down-regulate glucose transporter expression that correlates with increased oxidative stress in placental trophoblast cells in vitro. J Soc Gynecol Investig. 2004 Feb;11(2):75-81. doi: 10.1016/j.jsgi.2003.08.002. PMID 14980308
- [Background] von Lewinski D, Rainer PP, Gasser R, Huber MS, Khafaga M, Wilhelm B, Haas T, Machler H, Rossl U, Pieske B. Glucose-transporter-mediated positive inotropic effects in human myocardium of diabetic and nondiabetic patients. Metabolism. 2010 Jul;59(7):1020-8. doi: 10.1016/j.metabol.2009.10.025. Epub 2009 Dec 31. PMID 20045149
- [Background] Bays H. From victim to ally: the kidney as an emerging target for the treatment of diabetes mellitus. Curr Med Res Opin. 2009 Mar;25(3):671-81. doi: 10.1185/03007990802710422. PMID 19232040
- [Background] Chao EC, Henry RR. SGLT2 inhibition--a novel strategy for diabetes treatment. Nat Rev Drug Discov. 2010 Jul;9(7):551-9. doi: 10.1038/nrd3180. Epub 2010 May 28. PMID 20508640
- [Background] Takata K. Glucose transporters in the transepithelial transport of glucose. J Electron Microsc (Tokyo). 1996 Aug;45(4):275-84. doi: 10.1093/oxfordjournals.jmicro.a023443. PMID 8888584
- [Background] Ferrannini E, Solini A. SGLT2 inhibition in diabetes mellitus: rationale and clinical prospects. Nat Rev Endocrinol. 2012 Feb 7;8(8):495-502. doi: 10.1038/nrendo.2011.243. PMID 22310849
- [Background] Polidori D, Sha S, Mudaliar S, Ciaraldi TP, Ghosh A, Vaccaro N, Farrell K, Rothenberg P, Henry RR. Canagliflozin lowers postprandial glucose and insulin by delaying intestinal glucose absorption in addition to increasing urinary glucose excretion: results of a randomized, placebo-controlled study. Diabetes Care. 2013 Aug;36(8):2154-61. doi: 10.2337/dc12-2391. Epub 2013 Feb 14. PMID 23412078
- [Background] Han S, Hagan DL, Taylor JR, Xin L, Meng W, Biller SA, Wetterau JR, Washburn WN, Whaley JM. Dapagliflozin, a selective SGLT2 inhibitor, improves glucose homeostasis in normal and diabetic rats. Diabetes. 2008 Jun;57(6):1723-9. doi: 10.2337/db07-1472. Epub 2008 Mar 20. PMID 18356408
- [Background] Rossetti L, Smith D, Shulman GI, Papachristou D, DeFronzo RA. Correction of hyperglycemia with phlorizin normalizes tissue sensitivity to insulin in diabetic rats. J Clin Invest. 1987 May;79(5):1510-5. doi: 10.1172/JCI112981. PMID 3571496
- [Background] McCrimmon RJ, Evans ML, Jacob RJ, Fan X, Zhu Y, Shulman GI, Sherwin RS. AICAR and phlorizin reverse the hypoglycemia-specific defect in glucagon secretion in the diabetic BB rat. Am J Physiol Endocrinol Metab. 2002 Nov;283(5):E1076-83. doi: 10.1152/ajpendo.00195.2002. PMID 12376337
- [Background] Yale JF, Bakris G, Cariou B, Yue D, David-Neto E, Xi L, Figueroa K, Wajs E, Usiskin K, Meininger G. Efficacy and safety of canagliflozin in subjects with type 2 diabetes and chronic kidney disease. Diabetes Obes Metab. 2013 May;15(5):463-73. doi: 10.1111/dom.12090. Epub 2013 Mar 28. PMID 23464594
- [Background] Stenlof K, Cefalu WT, Kim KA, Alba M, Usiskin K, Tong C, Canovatchel W, Meininger G. Efficacy and safety of canagliflozin monotherapy in subjects with type 2 diabetes mellitus inadequately controlled with diet and exercise. Diabetes Obes Metab. 2013 Apr;15(4):372-82. doi: 10.1111/dom.12054. Epub 2013 Jan 24. PMID 23279307
- [Background] Stenlof K, Cefalu WT, Kim KA, Jodar E, Alba M, Edwards R, Tong C, Canovatchel W, Meininger G. Long-term efficacy and safety of canagliflozin monotherapy in patients with type 2 diabetes inadequately controlled with diet and exercise: findings from the 52-week CANTATA-M study. Curr Med Res Opin. 2014 Feb;30(2):163-75. doi: 10.1185/03007995.2013.850066. Epub 2013 Oct 28. PMID 24073995
- [Background] Rosenstock J, Aggarwal N, Polidori D, Zhao Y, Arbit D, Usiskin K, Capuano G, Canovatchel W; Canagliflozin DIA 2001 Study Group. Dose-ranging effects of canagliflozin, a sodium-glucose cotransporter 2 inhibitor, as add-on to metformin in subjects with type 2 diabetes. Diabetes Care. 2012 Jun;35(6):1232-8. doi: 10.2337/dc11-1926. Epub 2012 Apr 9. PMID 22492586
- [Background] Schernthaner G, Gross JL, Rosenstock J, Guarisco M, Fu M, Yee J, Kawaguchi M, Canovatchel W, Meininger G. Canagliflozin compared with sitagliptin for patients with type 2 diabetes who do not have adequate glycemic control with metformin plus sulfonylurea: a 52-week randomized trial. Diabetes Care. 2013 Sep;36(9):2508-15. doi: 10.2337/dc12-2491. Epub 2013 Apr 5. PMID 23564919
- [Background] Lavalle-Gonzalez FJ, Januszewicz A, Davidson J, Tong C, Qiu R, Canovatchel W, Meininger G. Efficacy and safety of canagliflozin compared with placebo and sitagliptin in patients with type 2 diabetes on background metformin monotherapy: a randomised trial. Diabetologia. 2013 Dec;56(12):2582-92. doi: 10.1007/s00125-013-3039-1. Epub 2013 Sep 13. PMID 24026211
- [Background] Brady EM, Davies MJ, Gray LJ, Saeed MA, Smith D, Hanif W, Khunti K. A randomized controlled trial comparing the GLP-1 receptor agonist liraglutide to a sulphonylurea as add on to metformin in patients with established type 2 diabetes during Ramadan: the Treat 4 Ramadan Trial. Diabetes Obes Metab. 2014 Jun;16(6):527-36. doi: 10.1111/dom.12249. Epub 2014 Jan 26. PMID 24373063
- [Background] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542
- [Background] He YL, Foteinos G, Neelakantham S, Mattapalli D, Kulmatycki K, Forst T, Taylor A. Differential effects of vildagliptin and glimepiride on glucose fluctuations in patients with type 2 diabetes mellitus assessed using continuous glucose monitoring. Diabetes Obes Metab. 2013 Dec;15(12):1111-9. doi: 10.1111/dom.12146. Epub 2013 Jul 14. PMID 23782529
- [Background] Ziaee V, Razaei M, Ahmadinejad Z, Shaikh H, Yousefi R, Yarmohammadi L, Bozorgi F, Behjati MJ. The changes of metabolic profile and weight during Ramadan fasting. Singapore Med J. 2006 May;47(5):409-14. PMID 16645692
- [Background] Siaw MY, Chew DE, Dalan R, Abdul Shakoor SA, Othman N, Choo CH, Shamsuri NH, Abdul Karim SN, Chan SY, Lee JY. Evaluating the Effect of Ramadan Fasting on Muslim Patients with Diabetes in relation to Use of Medication and Lifestyle Patterns: A Prospective Study. Int J Endocrinol. 2014;2014:308546. doi: 10.1155/2014/308546. Epub 2014 Nov 11. PMID 25435876
- [Background] Grant PM, Ryan CG, Tigbe WW, Granat MH. The validation of a novel activity monitor in the measurement of posture and motion during everyday activities. Br J Sports Med. 2006 Dec;40(12):992-7. doi: 10.1136/bjsm.2006.030262. Epub 2006 Sep 15. PMID 16980531
- [Background] Plasqui G, Westerterp KR. Physical activity assessment with accelerometers: an evaluation against doubly labeled water. Obesity (Silver Spring). 2007 Oct;15(10):2371-9. doi: 10.1038/oby.2007.281. PMID 17925461
- [Background] McClain JJ, Sisson SB, Tudor-Locke C. Actigraph accelerometer interinstrument reliability during free-living in adults. Med Sci Sports Exerc. 2007 Sep;39(9):1509-14. doi: 10.1249/mss.0b013e3180dc9954. PMID 17805082
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Erondu N, Desai M, Ways K, Meininger G. Diabetic Ketoacidosis and Related Events in the Canagliflozin Type 2 Diabetes Clinical Program. Diabetes Care. 2015 Sep;38(9):1680-6. doi: 10.2337/dc15-1251. Epub 2015 Jul 22. PMID 26203064
- [Background] Beshyah SA. Fasting During The Month of Ramadan For People with Diabetes: Medicine and Fiqh United at Last. Ibnosina Journal of Medicine and Biomedical Sciences; 1(2):58-60 (2009).
- [Background] Valentine V. The role of the Kidney and Sodium-Glucose Cotransporter-Inhibition in diabetes Management. Clinical Diabetes; 30(4):151-155 (2012).
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938